CLINICAL TRIAL: NCT03059407
Title: Impact of Animal Assisted Therapy on Quality, Completeness, and Patient and Parental Satisfaction in Children Undergoing Clinical Echocardiography
Brief Title: Impact of Therapy Dog Presence on Pediatric Echocardiogram
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00081186
Record Dates: First submitted 2017-02-17; First posted 2017-02-23 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Dog Therapy

STUDY DESIGN:
Intervention Model Description: Subjects will be assigned into one of three groups: 1) Canine assisted therapy only; 2) Canine assisted therapy plus standard distraction techniques; and 3) Standard distraction techniques only.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dog therapy only (Other): Canine assisted therapy only during echocardiogram
  Interventions: Behavioral: Dog therapy only
- Dog plus standard distraction tech (Other): Canine assisted therapy plus standard distraction techniques during echocardiogram
  Interventions: Behavioral: Dog plus standard distraction tech
- Standard distraction technique only (Other): Standard distraction techniques only during echocardiogram.
  Interventions: Behavioral: Standard distraction techniques only

INTERVENTIONS:
Behavioral: Dog therapy only — Canine assisted therapy only during echocardiogram
  Arms: Dog therapy only
Behavioral: Dog plus standard distraction tech — Canine assisted therapy plus standard distraction techniques during echo
  Arms: Dog plus standard distraction tech
Behavioral: Standard distraction techniques only — Standard distraction techniques (such as watching a movie) only during echocardiogram
  Arms: Standard distraction technique only

SUMMARY:
Young children with known or suspected heart disease frequently have difficulty cooperating with a clinically ordered echocardiogram. Current distraction techniques vary in efficacy. There have been no studies examining the use of animal assisted therapy to improve echocardiogram quality and completeness, as well as the patient/parent experience.

Hypotheses:

1. The presence and interaction of therapy dogs with young children undergoing echocardiography in a clinical setting will result in more complete and higher quality echocardiograms compared to standard distraction techniques.
2. Parents will report higher visit satisfaction scores and greater exam comfort for their children for echocardiograms performed with the aid of canine assisted therapy compared to use of standard distraction techniques.

Study Activities and Population Group:

Pilot Phase: Introduction of trained therapy dogs (approved by the Pets at Duke Therapy Program) for 10 echocardiograms to observe canine-patient interactions and determine best practices for inclusion of dog/handler team into the echocardiogram protocol.

Study Phase: 150 subjects ages will be selected from all children ages 1 to 5 years presenting for clinically ordered echocardiograms during the study time period. Subjects will be assigned into one of three groups: 1) Canine assisted therapy only; 2) Canine assisted therapy plus standard distraction techniques; and 3) Standard distraction techniques only. Echocardiography reviewers will be blinded to subject study group and will assign quality and completeness score based on validated criteria. Parental satisfaction will be assessed using validated survey tools.

Data analysis and risk/safety issues:

All subjects will be assigned a random subject ID, with the only link to PHI stored in a Duke Redcap database. Statistical testing will be performed with the assistance of Tracy Spears (biostatistician in DCRI) who has assisted with development of testing tools. There are no physical risks associated with the echocardiogram portion of the study, and very minimal risks with the therapy dog portion of the study. Please see "Pets at Duke" policy included in study documents. There is a potential loss of confidentiality, although the only link between subject ID and PHI will be stored in a Duke Recap database.

DETAILED DESCRIPTION:
Design and Procedures:

160 study subjects will be selected from all children 1 to 5 years of age presenting to the Duke University Pediatric Echocardiography Laboratory for a clinically ordered echocardiogram during the study period.

Duke University Hospital has an established program for pet therapy that includes bedside visits from trained and certified therapy dogs. At present, these dog-handler teams are certified as therapy dogs, and then fulfill additional certification requirements in order to be allowed into patient rooms. As this program and certification requirements are already established, this project would be able to liaison with the Pets at Duke program to provide suitable dog-handler teams for the study. Therapy dog certification requires passage of the AKC Good Citizen Test as well as instruction and certification through a recognized therapy dog program (including North Carolina Pet Partners, and Carolina Canines for Service). Currently, dogs (of any breed) that are certified as therapy dogs undergo evaluation by a team at Duke University and, if appropriate, are able to perform lobby visits (Level 2 dogs) or bed/patient room visits (Level 3 dogs). Only Level 3 dogs would be included in this study.

Data Collection:

* Subject demographics (age, ethnicity, gender, birth order, home ZIP code, city/rural designation)
* Presence and type of heart disease and interventions, if any
* Presence of a dog (breed to be specified) or other pet at home, exposure to other animals
* History of any traumatic canine experience (fears, bites)
* Presence of parental anxiety with dogs
* Completeness of echocardiogram based on existing protocol QA document
* Quality of echocardiogram (poor, average, good, excellent)
* Time required to perform echocardiogram
* Assessment of echocardiogram complexity (low, medium, high)
* Patient and parental/guardian comfort and satisfaction with echocardiogram experience
* Handler assessment of dog comfort throughout echocardiogram
* Handler assessment of quality of dog-subject interaction

Echocardiography Data Echocardiography completeness, quality, time and complexity will be assessed by either co-PI, who will be blinded to the subject group or presence of a dog during the echocardiogram.

* Echo completeness will be assessed using a numerical version of the existing protocol document used for QA
* Quality of the echocardiogram will be assessed using a qualitative scale derived from published pediatric echocardiography studies
* Time required to perform echocardiogram will be measured from time stamp on first image to time stamp on last image, automatically displayed for each echo.

Video Recording of Therapy Dog Interaction with Subject A video recording of the therapy dog interaction with the subject will be performed. This video review is part of a separate Duke University study investigating how therapy dogs behave around young children (Duke IACUC Protocol A112-14-05) and will not be analyzed as part of this study. It is likely that an image of the subject will be captured on the video, but none of the subject's protected health information or subject ID number will be included with the video. No video recordings will be released beyond the therapy dog analysis.

Timeline:

The study will be broken into 4 distinct phases:

1. Initial Phase (3 months): Medical team training and inclusion of study metrics into daily routine of the Duke University Hospital Pediatric Echocardiography Laboratory.
2. Pilot phase (3 months):

   1. 10 non-randomized subjects will be recruited and matched with dog-handler teams
   2. Through observation of dog-handler-child behavior and suggested interventions, a list of techniques will be developed for use in the main study. This will be an extension of knowledge gained from patient visits performed by therapy dogs in other settings within Duke Hospital.

   i. Suggested interventions may include, but are not limited to: having the dog lie next to the child on the bed, having the child practice resting their hand on the dog, demonstrating probe placement on the dog prior to placement on the child c. The behaviors rated as most helpful by sonographers and dog handlers will be selected as a list of techniques from which to select for consistent use during the main study.
3. Study phase (12 months)

   1. Subjects will be approached for participation and randomized into study group as outlined above
   2. Study data will be collected as outlined above
4. Data analysis and manuscript submission (12 months)

ELIGIBILITY:
Inclusion Criteria:

* Study subjects will be selected from all children 1 to 5 years of age presenting to the Duke University Pediatric Echocardiography Laboratory (Duke Peds Echo Lab) for a clinically ordered echocardiogram during the study time period

Exclusion Criteria:

* parental or child refusal to participate;
* known allergy to dogs;
* fear of dogs;
* concern for overly aggressive child behavior towards the dog;
* or concern for immune system function/infectious risk that could be worsened by animal exposure.

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 138 (Actual)
Dates: Start 2017-05-25 (Actual); Primary Completion 2024-06-27 (Actual); Study Completion 2024-06-27 (Actual)

PRIMARY OUTCOMES:
Quality of echocardiogram | 1 hour
  Echocardiography completeness, quality, time and complexity will be assessed by co-PI, who will be blinded to the subject group or presence of a dog during the echocardiogram.

SECONDARY OUTCOMES:
Parent satisfaction | 1 hour
  This outcome will be measured by parent questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Piers Barker, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No